CLINICAL TRIAL: NCT02249117
Title: Pharmacokinetics and Pharmacodynamics of BIWH 3: a Randomised, Placebo-controlled, Double Blind Dose Escalation Study (0.02, 0.06, 0.2, 0.6, and 2.0 μg/kg Intravenous Over One Hour) in Healthy Duffy Positive vs. Duffy Negative Male Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of BIWH 3 in Healthy Duffy Positive vs. Duffy Negative Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1181.2
Record Dates: First submitted 2014-08-21; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BIWH 3 (Experimental): single escalating dose
  Interventions: Drug: BIWH 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIWH 3
  Arms: BIWH 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to compare the pharmacokinetic and pharmacodynamic effects of escalating dosages of recombinant human pyro-Glu MCP-1 (BIWH 3) in Duffy positive vs. Duffy negative healthy male volunteers: plasma levels of monocyte chemotactic protein-1 (MCP-1) and markers of leukocyte, coagulation, platelet and endothelial activation will be quantified; To examine the safety of BIWH 3 in this setting

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Erythrocyte Fy positive and negative individuals because expression of the Duffy (Fy) receptor may influence MCP-1 plasma levels in humans
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age ≥ 18 and ≤ 50 years
* Body mass index: ≥18 kg/m2 and < 30 kg/m2
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory variables unless the investigator considers an abnormality to be clinically irrelevant
* Normal pharmacodynamic variables as determined at baseline visit
* Normal response to glucose tolerance test

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Current or history of: gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, autoimmune, hormonal disorders, diseases of the central nervous system (such as epilepsy), psychiatric disorders or cancer
* Symptoms of a clinically relevant illness in the 3 weeks prior to planned administration of study drug
* History of orthostatic hypotension, fainting spells and blackouts
* Chronic or relevant acute infections
* History of allergy / hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Any Electrocardiogram (ECG) value outside the reference range of clinical relevance including, but not limited to QRS interval > 110 ms or QTcB > 450 ms
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to planned administration of study drug
* Use of any drugs which might influence the results of the trial within 10 days prior to planned administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to planned administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Current or history of drug, alcohol, tobacco or caffeine abuse
* Blood donation within 1 month prior to planned administration or during the trial
* Excessive physical activities within 5 days prior to planned administration of study drug or during the trial
* Seropositivity for hepatitis B antigen (HBs-Ag), hepatitis C (HCV), HIV 1, or HIV 2 antibodies
* Weight over 95 kg

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2003-06; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve extrapolated to infinity (AUC0-∞) | up to 14 days after drug administration
Area under the plasma concentration-time curve up to the last quantifiable plasma concentration (AUC0-tz) | up to 14 days after drug administration
maximum BIWH 3 plasma concentration (Cmax) | up to 14 days after drug administration

SECONDARY OUTCOMES:
Monocyte activation | up to 14 days after drug administration
  Quantification of leukocyte surface markers by flow cytometry
Platelet cell activation | up to 14 days after drug administration
  Quantification of soluble P-selectin by enzyme immunoassay
Endothelial cell activation | up to 14 days after drug administration
  Quantification of soluble E-selectin by enzyme immunoassay
Inflammatory response | up to 14 days after drug administration
  Quantification of mRNA expression of IL-1 by reverse transcriptase-polymerase chain reaction (RT-PCR)
Activation of coagulation | up to 14 days after drug administration
  Prothrombin fragment levels via an enzyme-immunoassay
Number of subjects with adverse events | up to 14 days after drug administration
Number of subjects with clinically significant findings in vital signs | up to 14 days after drug administration
  blood pressure, pulse rate, body temperature
Number of subjects with clinically significant findings in ECG | up to 14 days after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 14 days after drug administration